CLINICAL TRIAL: NCT05914727
Title: Biomarkers Of Lung InVolvement In ASMD
Acronym: BOLIVIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eline C. B. Eskes (Other)
Responsible Party: Sponsor-Investigator, Eline C. B. Eskes, MD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020_298#B2021154
Record Dates: First submitted 2023-06-06; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Asmd, Visceral Type
MeSH Terms: conditions — Niemann-Pick Disease, Type B

STUDY DESIGN:
Intervention Model Description: This study comprises a cross-sectional case-control part and a prospective cohort part. In the cross-sectional part, exhaled breath samples with volatile and non-volatile compounds of ASMD patients and healthy controls will be collected. After potential biomarkers are identified in the cross-sectional part, patients will enter the longitudinal part in which the prognostic and monitoring value of these markers will be evaluated using clinical parameters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASMD patients (Other): ASMD patients
  Interventions: Diagnostic Test: eNose; Diagnostic Test: Volatile exhaled breath sample; Diagnostic Test: Condensate sample
- Healthy controls (Other): Healthy controls
  Interventions: Diagnostic Test: eNose; Diagnostic Test: Volatile exhaled breath sample; Diagnostic Test: Condensate sample

INTERVENTIONS:
Diagnostic Test: eNose — Collection of breath profile with eNose
Diagnostic Test: Volatile exhaled breath sample — Collection of exhaled breath in Tedlar bag
Diagnostic Test: Condensate sample — Collection of exhaled breath condensate with EcoScreen

SUMMARY:
The goal of this study is to characterize ASMD patients' breath profile, exhaled breath and condensate as compared to healthy controls to identify specific volatile and non-volatile compounds that reflect inflammatory processes, fibrotic processes or sphingolipid accumulation in the lungs.

Participants will be provided exhaled breath samples in three ways (breath profile, volatile compounds and condensate). ASMD patients will be compared to age- and sex-matched healthy controls.

DETAILED DESCRIPTION:
Rationale: Acid sphingomyelinase deficiency (ASMD) is a lysosomal storage disease in which sphingomyelin accumulates due to a deficiency of the enzyme acid sphingomyelinase. The most common manifestations of the chronic visceral subtype of this disease are hepatosplenomegaly and interstitial lung disease (ILD). Currently, enzyme replacement therapy is under investigation and will likely become available in the near future. The first results indicate that pulmonary involvement may be responsive to treatment. In order to identify those patients that will potentially benefit from therapy, biomarkers for lung injury can be helpful. Compounds measured in exhaled breath and exhaled breath condensate are extensively studied in common lung diseases and increasingly in ILD. These compounds are of interest since they provide information directly form the lung compartment and are collected non-invasively.

Objective: Our aim is to characterize ASMD patients' breath profile, exhaled breath and condensate as compared to healthy controls to identify specific volatile and non-volatile compounds that reflect inflammatory processes, fibrotic processes or sphingolipid accumulation in the lungs.

Study design: This study comprises a cross-sectional case-control part and a prospective cohort part. In the cross-sectional part, exhaled breath samples with volatile and non-volatile compounds of ASMD patients and healthy controls will be collected. After potential biomarkers are identified in the cross-sectional part, patients will enter the longitudinal part in which the prognostic and monitoring value of these markers will be evaluated using clinical parameters.

Study population: ASMD patients ≥ 12 years of age with a confirmed diagnosis of the chronic visceral type will be included as well as age-, sex- and smoking status-matched healthy controls with a ratio of 1:3.

Main study parameters/endpoints: Inflammatory markers, fibrotic markers and markers of sphingolipid accumulation will be measured in exhaled breath. Breath profiles will be measured with eNose, volatile compounds will be measured with GC-MS and non-volatile compounds will be measured in exhaled breath condensates using UPLC-MS/MS.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Sampling of exhaled breath yields no risk: at most, patients might suffer from dizziness or mild dyspnea. Patients will not directly benefit from participation in the study. We aim to identify biomarkers reflecting lung involvement of ASMD and in that respect the results of the study may improve clinical care in the future for the patients participating in the study or any ASMD patient with similar characteristics.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* The patient has a biochemical and genetically confirmed diagnosis of the chronic visceral subtype of ASMD
* The patient is willing and able to provide written informed consent prior to the study-related procedure.
* The patient is ≥ 12 years of age

Healthy controls:

* The individual is willing and able to provide written informed consent prior to the study-related procedure
* The individual is ≥ 16 years of age
* General good health as determined by medical history

Exclusion Criteria:

Patients:

* Inability to adhere to the study protocol
* When a patient is not able to complete a spirometry test, the eNose sample will not be collected.

Healthy controls:

* Medical history of (systemic) disease for which medication was necessary
* Inability to adhere to the study protocol

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Markers of inflammation, fibrosis or sphingolipid accumulation in exhaled breath | 1 year
  Markers of inflammation, fibrosis or sphingolipid accumulation in exhaled breath of ASMD patients. Since this is an explorative study these markers cannot be defined in advance.

SECONDARY OUTCOMES:
Biomarkers with monitoring or prognostic value in ASMD | 10 years
  Biomarkers with monitoring or prognostic value in ASMD patients in a longitudinal study design. Since this is an explorative study these markers cannot be defined in advance.

CONTACTS AND LOCATIONS:
Overall Officials: Carla EM Hollak, MD, PhD, prof, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Research data will be submitted as articles to peer-reviewed journals. Also, an abstract of our research data reporting our findings will be submitted for presentations on scientific, public and/or patient organization meetings for oral presentation(s).